CLINICAL TRIAL: NCT06031441
Title: A Phase I, Open-Label, Multicenter, Dose-Escalation Study Evaluating the Safety, Pharmacokinetics, and Activity of RO7566802 as a Single Agent and in Combination With Atezolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Activity of RO7566802 as a Single Agent and in Combination With Atezolizumab in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO44431; 2023-509266-38-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Solid Tumors; Recurrent Solid Tumors; Metastatic Solid Tumors
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Participants in successive cohorts will receive escalating doses of RO7566802, as an intravenous (IV) infusion on Day 1 of each 21-day cycle followed by RO7566802 in combination with a fixed dose of atezolizumab, as an IV infusion on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO7566802; Drug: Atezolizumab
- Dose Expansion Cohort (Experimental): Participants with select solid tumors will receive a recommended dose of RO7566802, determined in Dose Escalation phase, as an IV infusion in combination with a fixed dose of atezolizumab, as an IV infusion on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: RO7566802; Drug: Atezolizumab

INTERVENTIONS:
Drug: RO7566802 — RO7566802 solution for infusion will be administered as specified in each treatment arm.
Drug: Atezolizumab — Atezolizumab solution for infusion will be administered as specified in each treatment arm.
  Other Names: Tecentriq®

SUMMARY:
This is a first-in-human Phase I, open-label, dose-escalation and expansion study designed to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, pharmacodynamic, and preliminary anti-tumor activity of RO7566802 as a single agent and in combination with atezolizumab in participants with locally advanced, recurrent, or metastatic incurable solid tumor malignancies. Participants will be enrolled in 2 stages: dose escalation and expansion.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life expectancy >=3 months, in the investigator's judgment
* Adequate hematologic and end-organ function
* Histologically confirmed locally advanced, recurrent, or metastatic incurable solid tumor malignancy that has progressed after available standard therapy; or for whom standard therapy has proven to be ineffective or intolerable or is considered inappropriate; or for whom a clinical trial of an investigational agent is a recognized standard of care
* Measurable disease per RECIST v1.1
* Tumor specimen availability, for certain cohorts

Exclusion Criteria:

* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to Cycle 1 Day 1, with certain exceptions
* Active hepatitis B or C
* Active tuberculosis
* Positive test for human immunodeficiency virus (HIV) infection
* Administration of a live, attenuated vaccine (e.g., Flumist) within 4 weeks prior to RO7566802 infusion
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Active or history of autoimmune disease
* Prior allogeneic stem cell or organ transplantation
* Uncontrolled tumor-related pain
* Significant cardiovascular disease

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicity (DLTs) | Cycle 1 Day 1 through 21 days after Cycle 2 Day 1 (Cycle length=21 days) (up to approximately 42 days)
Percentage of Participants with Adverse Events (AEs) Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0) | Up to approximately 4 years

SECONDARY OUTCOMES:
Area Under the Serum Concentration Time Curve (AUC) of RO7566802 | Up to approximately 4 years
Maximum Serum Concentration (Cmax) of RO7566802 | Up to approximately 4 years
Minimum Serum Concentration (Cmin) of RO7566802 | Up to approximately 4 years
Total Clearance (CL) of RO7566802 | Up to approximately 4 years
Volume of Distribution at Steady State (Vss) of RO7566802 | Up to approximately 4 years
Serum Concentration of Atezolizumab | Up to approximately 4 years
Objective Response Rate as Determined by Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Up to approximately 4 years
Percentage of Participants with Anti-Drug Antibodies (ADAs) to RO7566802 | From Baseline up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- United States (6):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Yale Cancer Center, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai (ISMMS), New York, New York
  - The Ohio State University, Columbus, Ohio
  - Magee-Woman's Hospital, Harrisburg, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- Canada (2):
  - British Columbia Cancer Agency - 600 10th Ave W, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- United Kingdom (6):
  - Addenbrooke's Hospital, Cambridge
  - Leicester Royal Infirmary, Leicester
  - St Bartholomew's Hospital, London
  - Sarah Cannon Research Institute, London
  - Churchill Hospital, Oxford
  - The Royal Marsden hospital, Sutton

IPD SHARING:
Plan to Share IPD: No